CLINICAL TRIAL: NCT01459068
Title: Study of Effectiveness of Mental Health Interventions Among Torture Survivors on the Thailand-Burma Border
Brief Title: Mental Health Assessment Project on the Thailand-Burma Border
Acronym: MHAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Burma Border Projects (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00003601; DFD-A-00-08-00308-0 (Other: USAID)
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Depression; Anxiety; Posttraumatic Stress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waitlist-Control (No Intervention): Eligible study subjects were assigned to the waitlist-control arm on a rolling admissions basis. The waitlist-controls waited for a period equivalent to the duration of the intervention and then were re-interviewed.
- Common Elements Treatment Approach (Experimental): Eligible study subjects randomized into the CETA intervention were offered ten weeks of counseling sessions, consisting of nine elements designed to treat symptoms of common mental health disorders including depression, PTS, and anxiety and to provide skills to deal with life stressors.
  Interventions: Behavioral: Common Elements Treatment Approach

INTERVENTIONS:
Behavioral: Common Elements Treatment Approach — CETA components include:
  1. Engagement (encouraging participation)
  2. Psychoeducation (introduction)
  3. Anxiety Management Strategies (relaxation)
  4. Behavioral Activation (getting active)
  5. Cognitive Coping/Restructuring (thinking in a different way, part I and part II)
  6. Imaginal Gradual Exposure (talking about difficult memories)
  7. In Vivo Exposure (Live exposure)
  8. Suicide/Homicide/Danger Assessment and Planning (safety)
  9. Screening and Brief Intervention for Alcohol (alcohol intervention)
  Other Names: CETA
  Arms: Common Elements Treatment Approach

SUMMARY:
The aim of the study is to determine the effectiveness of a transdiagnostic psychotherapy intervention - namely, Common Elements Treatment Approach (CETA) - in reducing the severity of mental health symptoms experienced by torture and violence survivors displaced from Burma into Thailand. Specifically, the intervention seeks to measure reductions (if any) in symptoms of depression and trauma.

DETAILED DESCRIPTION:
The study is part of an award by the USAID Victims of Torture Fund (USAID/VTF) to JHU to work with local and international organizations serving survivors of torture and systematic violence. For this study, the intent is to assist in the design, implementation, monitoring, and evaluation of programming to understand and address the psychosocial needs of Burmese displaced across the Thai/Burma border who are living in the area of Mae Sot, Tak Province in Thailand. Specifically this project involves collaboration with the Burma Border Projects (BBP), the Mae Tao Clinic (MTC), the Assistance Association for Political Prisoners (AAPP), and Social Action for Women (SAW), to help improve the quality and effectiveness of psychosocial and mental health programs.

The Common Elements Treatment Approach (CETA) is a transdiagnostic treatment approach developed for delivery by lay counselors in low and middle income countries (LMIC) with few mental health professionals. CETA was designed to treat symptoms of common mental health disorders including depression, PTS, and anxiety, and to provide skills to deal with life stressors. includes engagement, psychoeducation, anxiety management strategies, behavioral activation, cognitive coping/restructuring, imaginal gradual exposure, suicide/homicide/danger assessment and planning, and screening and brief intervention for alcohol.

ELIGIBILITY:
Inclusion Criteria:

* Burmese national, 18 or over, living in Thailand outside of refugee camps, meets or exceed the algorithm for the Hopkins Symptoms Checklist 25 (HSCL-25) depression subscale and/or the algorithm for the Harvard Trauma Questionnaire (HTQ) posttraumatic stress scale.

Exclusion Criteria:

* not Burmese national, under 18, not living in Thailand outside of refugee camps, does not meet meet or exceed the algorithm for the Hopkins Symptoms Checklist 25 (HSCL-25) depression subscale and/or the algorithm for the Harvard Trauma Questionnaire (HTQ) posttraumatic stress scale; active psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtland Robinson, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Assistance Association for Political Prisoners; Mae Tao Clinic; Social Action for Women, Mae Sot, Changwat Tak, Thailand

REFERENCES:
- [Derived] Bolton P, Lee C, Haroz EE, Murray L, Dorsey S, Robinson C, Ugueto AM, Bass J. A transdiagnostic community-based mental health treatment for comorbid disorders: development and outcomes of a randomized controlled trial among Burmese refugees in Thailand. PLoS Med. 2014 Nov 11;11(11):e1001757. doi: 10.1371/journal.pmed.1001757. eCollection 2014 Nov. PMID 25386945

RESULTS

PARTICIPANT FLOW:
Groups:
- Common Elements Treatment Approach: Eligible study subjects randomized into the CETA intervention were offered ten weeks of counseling sessions, consisting of nine elements designed to treat symptoms of common mental health disorders including depression, PTS, and anxiety and to provide skills to deal with life stressors.
  Common Elements Treatment Approach: CETA components include:
  1. Engagement (encouraging participation)
  2. Psychoeducation (introduction)
  3. Anxiety Management Strategies (relaxation)
  4. Behavioral Activation (getting active)
  5. Cognitive Coping/Restructuring (thinking in a different way, part I and part II)
  6. Imaginal Gradual Exposure (talking about difficult memories)
  7. In Vivo Exposure (Live exposure)
  8. Suicide/Homicide/Danger Assessment and Planning (safety)
  9. Screening and Brief Intervention for Alcohol (alcohol intervention)
Period: Overall Study
Arm/Group | Waitlist-Control | Common Elements Treatment Approach
Started | 165 | 182
Completed | 126 | 148
Not Completed | 39 | 34
Not completed — Withdrawal by Subject | 8 | 18
Not completed — Lost to Follow-up | 31 | 15
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: We estimated 150 participants in each arm using the test for paired means, based on a moderate effect size (0.50), 80% power, two-tailed 5% significance level, design effect of 1.5, and up to a 50% expected drop-out rate (due to frequent cross-border movement).
Groups:
- Total: Total of all reporting groups
Arm/Group | Waitlist-Control | Common Elements Treatment Approach | Total
Number analyzed (Participants) | 165 | 182 | 347
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (11.4) | 36.5 (12.6) | 35.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 111 | 217
  Male | 59 | 71 | 130

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: Depression symptoms were measured using a modified, locally validated version of the 15-item Hopkins Symptoms Checklist (HSCL-25) depression subscale. Respondents reported symptom frequency in the last month (0 "None of the time" to 3 "Almost always"). An algorithm was applied to the HSCL-25 to determine eligibility on the basis of moderate to severe depression. The HSCL-25 was also used to measure the depression severity outcome: Scores on the depression scale were calculated as average symptom scores across the 17 items and therefore ranged from 0-3
Time Frame: 10-16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Waitlist-Control | Common Elements Treatment Approach
Number analyzed (Participants) | 165 | 182
units on a scale | -0.52 (.06) | -1.02 (.05)
Statistical Analysis 1: Comparison: Waitlist-Control vs Common Elements Treatment Approach; Test type: Non-Inferiority or Equivalence — We estimated 150 participants in each arm using the test for paired means, based on a moderate effect size (0.50), 80% power, two-tailed 5% significance level, design effect of 1.5, and up to a 50% expected drop-out rate (due to frequent cross-border movement); p < 0.001, longitudinal model — a priori threshold for statistical significance was 0.05; longitudinal to model within-person change in mean scores; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.59 to -0.40], Standard Error of Mean .05

2. Secondary Outcome: Functional Impairment
Description: Functional impairment was measured using locally-developed, gender-specific scales. The scales contained 16 and 23 tasks for men and women, respectively. Respondents reported current difficulty compared to others of same gender and similar age (from 0 "No difficulty" to 4 "Often cannot do"). Scores were calculated as average task scores across the 16- and 23-item scales and therefore ranged from 0-4
Time Frame: 10-16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Waitlist-Control | Common Elements Treatment Approach
Number analyzed (Participants) | 165 | 182
units on a scale | -0.20 (.09) | -0.64 (.10)
Statistical Analysis 1: Comparison: Waitlist-Control vs Common Elements Treatment Approach; Test type: Non-Inferiority or Equivalence — power calculations were not done for secondary outcomes; p < 0.001, longitudinal model; Mean Difference (Net) = -0.44, 95% CI 2-sided [-0.59 to -0.28], Standard Error of Mean .10

3. Primary Outcome: Posttraumatic Stress Symptoms
Description: Posttraumatic stress symptoms (PTSS) were measured using the 30-symptom items of the Harvard Trauma Questionnaire (HTQ). Response options were the same as the HSCL-25. An algorithm was applied to the HTQ to determine eligibility on the basis of moderate to severe PTSS. The HTQ was also used to measure the PTSS severity outcome: Scores for PTSS were calculated as average symptom scores across the 30 items. PTSS scores ranged from 0 (best possible outcome) to 3 (worst possible outcome).
Time Frame: 10-16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Waitlist-Control | Common Elements Treatment Approach
Number analyzed (Participants) | 165 | 182
units on a scale | -0.38 (.05) | -0.80 (.04)
Statistical Analysis 1: Comparison: Waitlist-Control vs Common Elements Treatment Approach; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, longitudinal model — a priori threshold for significance set at 0.05; longitudinal analysis modeling within-person change in mean scores; Mean Difference (Net) = -0.43, 95% CI 2-sided [-0.51 to -0.35], Standard Error of Mean 0.04

4. Secondary Outcome: Anxiety Symptoms
Description: Anxiety symptoms were measured using the 10-item HSCL-25 anxiety subscale with local adaptations. Respondent instructions and response categories were the same as the HSCL-25 depression subscale. Scores were calculated as average symptom scores across the 11-item scale and therefore ranged from 0-4
Time Frame: 10-16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Waitlist-Control | Common Elements Treatment Approach
Number analyzed (Participants) | 165 | 182
units on a scale | -0.42 (0.09) | -0.90 (0.08)
Statistical Analysis 1: Comparison: Waitlist-Control vs Common Elements Treatment Approach; Test type: Non-Inferiority or Equivalence — no power calculations on secondary outcomes; p < 0.001, longitudinal model; Mean Difference (Net) = -0.48, 95% CI 2-sided [-0.61 to -0.34], Standard Error of Mean 0.07

5. Secondary Outcome: Aggression Behaviors
Description: The 12-item Aggression Questionnaire (AQ) was adapted for local use. Respondents rated frequency in general of aggressive behaviors from 0 "None of the time" to 4 "Almost all of the time." Scores were calculated as averages scores for each behavior across the 12-item scale and therefore ranged from 0-4
Time Frame: 10-16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Waitlist-Control | Common Elements Treatment Approach
Number analyzed (Participants) | 165 | 182
units on a scale | -0.22 (0.05) | -0.47 (0.03)
Statistical Analysis 1: Comparison: Waitlist-Control vs Common Elements Treatment Approach; Test type: Non-Inferiority or Equivalence — no power calculations for secondary measures; p < 0.001, longitudinal model; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.34 to -0.15], Standard Error of Mean 0.05

6. Secondary Outcome: Alcohol Use
Description: Alcohol use was measured using the Alcohol Use Disorders Identification Test (AUDIT). Respondents reported frequency and amount of alcohol consumed, referencing photographs of local alcohols (local beers, rice whiskeys, etc.). Total scores were calculated as sum totals across the 10-item scale. AUDIT total scores ranged from 0 (best possible outcome) to 40 (worst possible outcome).
Time Frame: 10-16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Waitlist-Control | Common Elements Treatment Approach
Number analyzed (Participants) | 15 | 18
units on a scale | -1.29 (0.21) | -1.25 (0.17)
Statistical Analysis 1: Comparison: Waitlist-Control vs Common Elements Treatment Approach; Test type: Non-Inferiority or Equivalence — no power calculations for secondary measures; p = 0.896, longitudinal model; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.44 to 0.50], Standard Error of Mean 0.26

ADVERSE EVENTS:
Arm/Group | Waitlist-Control | Common Elements Treatment Approach
Serious Adverse Events (participants affected / at risk) | 0/165 | 0/182
Other Adverse Events (participants affected / at risk) | 0/165 | 0/182

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No